CLINICAL TRIAL: NCT03011242
Title: DC-STAMP: Regulators of Osteoclastogenesis and Response Marker in PsA
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D.; M.P.H.; Professor of Medicine, Chief of Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB 60239; 1R01AR069000-01 (NIH)
Record Dates: First submitted 2016-09-20; First posted 2017-01-05 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; US; DC-STAMP; Osteoclast Precursor (OCPs)
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If patient consents, peripheral blood samples that remain after study assays are completed may be stored for future non-genetic research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Longitudinal Cohort: Psoriatic Arthritis: Individuals diagnosed with Psoriatic Arthritis starting standard of care treatment with a TNFi or non-biologic DMARD.
- Assay Development: Healthy or Psoriatic Arthritis: Individuals that are healthy or with a diagnosis of Psoriatic Arthritis will be enrolled for blood draws for assay development and/or for an ultrasound for development of techniques and scoring system validation.
- Cross-Sectional: Psoriatic Arthritis: Individuals diagnosed with Psoriatic Arthritis in good disease state on stable non-biologic DMARDS or on stable TNFi.

SUMMARY:
The Investigators will examine if DC-STAMP can serve as an early marker of TNFi response in PsA. Identification of such a biomarker would permit rapid transition to a new agent, a major treatment advance. TNFi are the most effective therapies in PsA, however, methotrexate is frequently initiated early in the disease course based on its significantly lower cost. Unfortunately, the efficacy of MTX has not been supported in clinical trials and up to 40% of patients do not respond to TNFi therapy. Moreover, valid biomarkers to predict MTX or TNFi responses are currently unavailable. This study may also provide the first data on the comparative efficacy of MTX and TNFi using clinical, Ultrasound (US) and biomarker outcomes.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA), an inflammatory joint disease associated with psoriasis (Ps), affects approximately 650,000 adults in the United States and is associated with increased morbidity and mortality. Bone damage develops in half these patients within the first two years of the disease, often leaving them with impaired function and diminished quality of life. The emergence of anti-Tumor Necrosis Factor therapies (TNFi) has dramatically improved clinical response and slowed bone and cartilage degradation in PsA patients, however, only 50-60% of patients respond to these agents. To improve these outcomes, the investigators must address two major gaps: a limited understanding of key events that underlie pathologic bone destruction and the absence of biomarkers to predict biologic response and identify early biologic responders to facilitate optimization of therapy.

Bone damage is mediated by osteoclasts which arise from monocyte precursors in the blood. Osteoclast Precursors (OCPs) are dramatically increased in PsA, compared to controls, particularly in patients with bone damage on X-ray. The number of these circulating precursor cells dropped rapidly following treatment with TNFi. OCPs may serve as response biomarkers, but cost, time and high variability limit these assays. Osteoclast precursors express Dendritic Cell-Specific Transmembrane Protein (DC-STAMP), which is a seven-pass transmembrane protein required for fusion of monocytes to form osteoclasts and giant cells. Monocyte DC-STAMP levels dropped rapidly following treatment with TNFi. TNF receptor-associated factor 3 (TRAF3), an inhibitor of OC formation that correlates with extracellular TNF concentrations, is elevated in OCPs from PsA patients. These markers may predict TNFi treatment response.

The goal of this study is to examine DC-STAMP in Psoriatic Arthritis patients prior to and after starting standard of care treatment with a TNFi or non-biologic DMARD. We will also examine PsA patients with low disease activity on standard of care TNFi and PsA patients with low disease activity on standard of care non-biologic DMARDs will serve as controls.

Three groups of subjects will be recruited.

1. Longitudinal: 30 subjects starting out on standard of care treatment with a TNFi or non-biologic DMARD will take part in the longitudinal section of the study. Subjects may be asked to have a blood draw at one additional visit before starting therapy for additional research assays if they are DC-STAMP positive. If the longitudinal subjects that return for an additional blood draw before starting medication have unusable sample data, they will be replaced by additional longitudinal subjects out of the 30 enrolled longitudinal participants to get sufficient data results of two subjects. The subjects with unusable data will continue in the longitudinal follow up study visits as intended.
2. Cross sectional: 36 patients will take part in the cross-sectional part of the study. 18 patients on stable non-biologic DMARDS and 18 patients on stable TNFi will be compared in the cross-sectional part. This population should be in good disease state such that their disease is controlled and treatment will not need to be changed. If longitudinal subjects fit the cross-sectional criteria and wish to participate, they will be re-consented for the cross-sectional part of the study.

   While 66 subjects will be studied in both the longitudinal and cross-sectional studies combined, up to 80 PsA subjects may be consented to allow for screen failures and to replace longitudinal subjects who withdraw or are lost to follow-up.
3. Assay Development: Up to 40 PsA or healthy subjects may be enrolled for blood draw for assay development and to test development of techniques for ultrasound comparison and scoring system validation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Subjects can be of either gender but must be at least 18 years old.
* Subjects with PsA should fulfill CASPAR criteria.

  * Longitudinal: Patients with active PsA who will be starting a TNFi or non-biologic DMARD treatment (Subjects starting non-biologic DMARDS can have their blood drawn within the first few days of starting therapy).
  * Additional Blood Draw: Positive DC-STAMP signal at baseline
  * Cross-Sectional: Patients on stable DMARDS or TNFi for more than 16 weeks.
  * Healthy Subjects: Healthy controls should have no active systemic disorders or inflammatory conditions that would confound the results of the study.

Exclusion Criteria:

* Unable to donate blood because of poor venous access or intolerance of phlebotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects that are 18 years old and older. Due to the demographic distribution of the disease the investigators expect all or nearly all subjects to be caucasian, however no subjects will be excluded based on race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Assessing the Change of DC-STAMP as an early TNFi response biomarker. | Baseline to 2 weeks of standard of care treatment
  The Investigators will analyze the change in DC-STAMP expression from baseline to 2 weeks using flow cytometry.

SECONDARY OUTCOMES:
Assessing the Change of Clinical Response at 16 weeks. | Baseline to 16 weeks of standard of care treatment
  The Investigators will measure clinical response from baseline to 16 weeks using the Disease Activity Index for Psoriatic Arthritis (DAPSA). The cutoff points for the classification of disease activity states for the DAPSA are:
  remission less than or equal to 4, low disease activity 4-14, moderate disease activity 14-28, high disease activity >28

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD/MPH, Principal Investigator — Univerisity of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Samples of any type collected at the University of Rochester may be shared with researchers at other institutions. Subjects will be made aware of this in the informed consent form.
Time Frame: Once a subject signs the consent form to allow for sharing, if any samples remain after all tests are completed, the samples will be stored for future research indefinitely or until the subject cancels consent to share.
Access Criteria: Investigators at other collaborating institutions may have access to leftover samples and data. Data will not include any information that is identifying.

REFERENCES:
- See also: URMC Allergy, Immunology & Rheumatology Clinical Trials — https://www.urmc.rochester.edu/medicine/allergy/patients-families/clinical-trials.aspx